CLINICAL TRIAL: NCT04391868
Title: PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, 3-WAY, 6-SEQUENCE CROSSOVER STUDY TO DEMONSTRATE BIOEQUIVALENCE OF SILDENAFIL ORALLY-DISINTEGRATING FILM 50 MG WITH OR WITHOUT WATER TO ORAL TABLET OF SILDENAFIL CITRATE (VIAGRA(Registered)) 50 MG UNDER FASTED CONDITION IN HEALTHY MALE PARTICIPANTS
Brief Title: A Bioequivalence Study of Sildenafil Citrate Orally-Disintegrating Film Dosage Form
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The project has been transferred to Viatris
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A1481340
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Healthy
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Viagra tablet (Active Comparator): Subjects receive a single dose of 50 mg Viagra tablet followed by plasma sampling for 14 hours.
  Interventions: Drug: Viagra Tablet
- Sildenafil citrate ODF without water (Experimental): Subjects receive a single dose of 50 mg sildenafil ODF without water followed by plasma sampling for 14 hours.
  Interventions: Drug: Sildenafil Citrate ODF
- Sildenafil citrate ODF with water (Experimental): Subjects receive a single dose of 50 mg sildenafil ODF with water followed by plasma sampling for 14 hours.
  Interventions: Drug: Sildenafil Citrate ODF

INTERVENTIONS:
Drug: Viagra Tablet — 50 mg tablet on Day 1 of each period
  Arms: Viagra tablet
Drug: Sildenafil Citrate ODF — 50 mg ODF on Day 1 of each period
  Arms: Sildenafil citrate ODF without water
Drug: Sildenafil Citrate ODF — 50 mg ODF on Day 1 of each period
  Arms: Sildenafil citrate ODF with water

SUMMARY:
The purpose of this study is to assess the bioequivalence of Sildenafil ODF 50 mg to Viagra® tablet 50 mg under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, gastric bypass).
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb or HCVAb. Hepatitis B vaccination is allowed.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Participants who are currently prescribed and/or taking nitrates or nitric oxide donors in any form on either a regular or intermittent basis.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * AST or ALT level ≥1.5 × ULN;
  * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is≤ ULN.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2021-04-28 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Maximum Observed Plasma Concentration (Cmax) | 0, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose
  Maximum Observed Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) by Seriousness and Relationship to Treatment | Baseline up to 2 days after last dose of study medication
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to 2 days after last dose of study medication
  Laboratory parameters included: hematology, chemistry and urine. Clinical significance of laboratory parameters was determined at the investigator's discretion.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 2 days after last dose of study medication
  Vital signs are obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings | Baseline up to 2 days after last dose of study medication
  Physical examination included examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings were considered to be clinically significant based on investigator's decision.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A1481340